CLINICAL TRIAL: NCT00546104
Title: A Phase II Trial of Dasatinib to Treat Women With Stage IV or Inoperable Stage III Advanced Breast Cancer
Brief Title: Phase II Dasatinib Study in Advanced Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007578; BMS CA180089
Record Dates: First submitted 2007-10-16; First posted 2007-10-18 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced Breast Cancer; Breast cancer; Dasatinib; Inoperable Stage III Breast Cancer; Metastatic Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dasatinib (Experimental): 50- 100 mg PO BID
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — An initial dose of 50 mg PO BID; following 4 weeks of treatment, dose adjustment will be based on inhibition of phosphorylation of FAK and paxillin per biopsy assessment, as well as toxicity assessment.
  Other Names: Sprycel; BMS-354825

SUMMARY:
The purpose of this study is to find out if dasatinib will safely reduce the size or spread of your tumor.

DETAILED DESCRIPTION:
The introduction of biologics with specific molecular targets has initiated a trend toward improved survival in women with metastatic breast cancer.

The tyrosine kinase SRC (pp60src) is a member of a family of proteins that contribute to cellular signal transduction activities such as cell growth, differentiation, survival, adhesion and migration. Abnormal signaling has been linked to cancer metastases; thus, identification of molecular regulators or inhibitors of SRC present therapeutic opportunity for cancer patients. Src kinases consist of eight non-receptor tyrosine kinases (Src, Fyn, Yes, Lck, Lyn, Hck, Fgr and Blk) that interact with the intracellular domains of growth factor/cytokine receptors, (G-protein-coupled receptor)GPCRs and integrins.

Inhibition of SRC has also been associated with reversal of chemoresistance and restored sensitivity to drug-resistant ovarian cancer cells, suggesting potential as second- line treatment for previously treated populations. Dasatinib is a potent, broad spectrum inhibitor of 5 critical oncogenic tyrosine kinases, including SRC.

Patients will receive dasatinib, a Src inhibitor, at an initial dose of 50 mg PO BID, with real-time PharmacoDynamic dose adjustment following 4 weeks of therapy based on inhibition of phosphorylation of SRC, focal adhesion kinase (FAK) and paxillin, until progression. The primary objective is to assess tolerability and estimate the proportion of patients who are progression-free at 16 weeks from the date of study enrollment.

A minimum of 2 (maximum of 3) tumor biopsies will be analyzed and compared for SRC signature: one at baseline (study enrollment, all patients); the second after 4 weeks of dasatinib therapy (all patients); and the third at progression (only patients who progress after a documented response).

Patients will receive continuous daily administration until documented disease progression, and will be followed until death.

The results of this study may be useful in designing future studies using dasatinib alone or in combination with chemotherapy, thus having the potential to alter the current standard of care in this incurable population.

Additional correlative studies will be conducted. Tumor biopsies will be analyzed and compared for SRC, pSRC, Ki67, and related genomic signatures.

ELIGIBILITY:
Inclusion Criteria:

* Measurable Stage IV or inoperable Stage III advanced breast cancer.
* There is no limit on the number of prior therapies.
* At least 3 weeks since prior chemotherapy, biological or hormonal therapy.
* At least 2 weeks since surgical biopsy.
* At least 3 weeks since major (open thoracic/abdominal/cardiac) surgery.
* No central nervous system (CNS) metastases except solitary brain metastasis
* No cardiac dysfunction
* left ventricular ejection fraction (LVEF) ≥ 50% as determined by multiple gated acquisition scan (MUGA)/echocardiogram
* Adequate blood counts
* Normal liver and kidney function
* Negative serum pregnancy test.
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or breast feeding.
* Prior treatment with dasatinib.
* Bone as the only site of disease.
* Significant gastrointestinal bleeding
* Septicemia, infection, acute hepatitis, hypokalemia, or hypomagnesemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-10; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Blackwell, MD, Principal Investigator — Duke University
Locations (3):
- United States (3):
  - Palm Beach Cancer Center Institute, West Palm Beach, Florida
  - Presbyterian Health Care, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be identified in cancer center outpatient clinics multi-site. The study will be introduced by a physician or caregiver known to the patient. We will need to review protected health information in order to identify subjects, and information resulting from this activity will be used only to assess eligibility of a subject.
Pre-assignment Details: Meds which inhibit platelet function/coagulation,potent inhibitors of cytochrome CYP3A, or meds that prolong the QT interval during study require a 7 day wash-out.IV bisphosphonates must be held for 2 wks before/6 wks after trial tx. Subjects must be 3 wks since prior to therapy, 2 wks since surgical bx and 3 wks since major surgery.
Groups:
- Dasatinib: 50-100 mg PO BID
Period: Overall Study
Arm/Group | Dasatinib
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Dasatinib: 50-100mg by mouth twice a day
Arm/Group | Dasatinib
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Estimation of the Proportion of Progression-free Patients at 16 Wks.
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or measurable increase in a non-target lesion, or the appearance of new lesions, or similar definition as appropriate.
  Proportion progression-free at 16 weeks.From first day of study related treatment with Dasatinib until the date of first documented progression or date of death from any cause, whichever came first.
Time Frame: 16 weeks
Population: 31 patients on this trial, 1 patient was found to have disease progression at 16-weeks, 16 patients had disease progression prior to 16 weeks, 8 patients were taken off-treatment due to toxicity, and 6 patients voluntarily withdrew from treatment. These latter two groups of patients were censored in the analysis of Progression Free Survival.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dasatinib: 50mg-100mg po BID
Arm/Group | Dasatinib
Number analyzed (Participants) | 31
percentage of participants | 0 [0 to 20]

2. Secondary Outcome: To Measure Response to Protocol Therapy Per RECIST Criteria
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression At least a 20% increase in the sum of the longest diameter (LD) of target lesions taking as a reference the smallest sum longest diameter recorded since treatment started, or the appearance of one or more new lesions.
  RECIST 1.0 Overall response:
  Complete Response (CR) Partial Response (PR) Stable Disease (SD) Progressive Disease (PD)
  CR= CR+CR and No new lesions PR= CR+SD; PR+SD and no new lesions SD= SD+SD and no new lesions PD= PD+any new lesions
Time Frame: 16 weeks
Population: Proportion with Best Response of Stable Disease
Measure: Number; unit: percentage of participants
Arm/Group | Dasatinib
Number analyzed (Participants) | 30
percentage of participants | 16.7

3. Secondary Outcome: Characterization and Comparison of SRC (A Protein Tyrosine Kinase)Dysregulation at Baseline (All Patients), After 4 Weeks of Dasatinib Treatment (All Patients), and at Progression (Only Patients Who Progress After Documented Response)
Description: For the 20 patients with evaluable biopsies at baseline and week 4, the median relative change from baseline in tissue biomarker levels of phospho-Src (p-Src)
Time Frame: 4 weeks
Population: Twenty patients with evaluable biopsies at baseline and 4 week follow-up
Measure: Median (Inter-Quartile Range); unit: percentage of change in p-SRC
Arm/Group | Dasatinib
Number analyzed (Participants) | 20
percentage of change in p-SRC | -0.125 [-0.41 to 0.153]
Statistical Analysis 1: Comparison: Dasatinib; The median change in SRC from baseline to 4 weeks was estimated; Test type: Superiority or Other; p = 0.3, t-test, 2 sided — The p-value is from a paired t-test to test the null hypothesis the mean relative change in Src from baseline to 4 weeks is equal to zero; Median Difference (Net) = -0.13, 95% CI 2-sided [-30 to 9], Standard Error of Mean 9

4. Secondary Outcome: Correlate SRC Dysregulation Results With Response to Dasatinib Therapy
Description: Since all patients progressed there is no comparison to between responders and non-responders.
Time Frame: 16 weeks
Population: 20 patients with baseline and 4 week Src measures. 11 patients came off due to screen failure, toxicity or progression before 4 week biopsy.
Measure: Mean (95% Confidence Interval); unit: percentage change in p-SRC
Arm/Group | Dasatinib
Number analyzed (Participants) | 20
percentage change in p-SRC | -.10 [-.30 to .10]
Statistical Analysis 1: Comparison: Dasatinib; Test type: Superiority or Other; p = 0.3, t-test, 1 sided; Median Difference (Net) = -.13, 95% CI 2-sided [-.30 to .10], Standard Error of Mean .10

5. Secondary Outcome: To Explore the Association Between Each Patient's SRC Signature and Their Time to Progression.
Description: Spearman's correlation between the change in SRC signature from baseline to 4 weeks and time to progression
Time Frame: Baseline Src measure to first progression
Population: 11 patients had both change in Src level and progression time intervals
Measure: Number; unit: correlation coefficient
Arm/Group | Dasatinib
Number analyzed (Participants) | 11
correlation coefficient | 0.27

6. Secondary Outcome: To Explore the Association Between Dasatinib and Osteoclastic Bone Resorption
Description: Not assessed secondary to limited number of subjects.
Time Frame: not assessed
Arm/Group | Dasatinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Dasatinib: 50-100mg po bid
Arm/Group | Dasatinib
Serious Adverse Events (participants affected / at risk) | 10/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dasatinib (N=31)
Pain (General disorders) | 2
Pain, back (General disorders) | 1
Pain, extrimity limb (General disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 1
Syncope (General disorders) | 1
Edema, limb (Blood and lymphatic system disorders) | 1
AST (Hepatobiliary disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pain, chest/thorax (General disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis (Blood and lymphatic system disorders) | 1
hyponatremia (General disorders) | 1
infection (Infections and infestations) | 1
diarrhea (Gastrointestinal disorders) | 1
fever (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dasatinib (N=31)
anorexia (General disorders) | 13 (13) — grade 1 19% grade 2 13% grade 3 10%
fatigue (General disorders) | 16 (16) — number of subject effected: Grade 1=7 grade 2=8 grade 3=1
fever: non-neutropenic (Gastrointestinal disorders) | 5 (5) — number of subjects effected: Grade 1=3 grade 2=2 grade 3=0
Flushing (General disorders) | 7 (7) — number of subjects effected: Grade 1=5 grade 2=2 grade 3=0
insomnia (General disorders) | 8 (8) — number of subjects effected: Grade 1=6 grade 2=2 grade 3=0
diarrhea (Gastrointestinal disorders) | 15 (15) — number of subjects effected: Grade 1=10 grade 2=5 grade 3=0
constipation (Gastrointestinal disorders) | 11 (11) — number of subjects effected: Grade 1=8 grade 2=3 grade 3=0
nausea (Gastrointestinal disorders) | 19 (19) — number of subjects effected: Grade 1=10 grade 2=8 grade 3=1
vomiting (Gastrointestinal disorders) | 13 (13) — number of subjects effected: Grade 1=10 grade 2=3 grade 3=0
cough (Respiratory, thoracic and mediastinal disorders) | 6 (6) — number of subjects effected: Grade 1=6 grade 2=0 grade 3=0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (12) — number of subjects effected: Grade 1=4 grade 2=5 grade 3=3
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) — number of subjects effected: Grade 1=0 grade 2=1 grade 3=2
paricardial effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — number of subjects effected: Grade 1=2 grade 2=0 grade 3=0
pain: abdomen (Gastrointestinal disorders) | 6 (6) — number of subjects effected: Grade 1=6 grade 2=0 grade 3=0
pain: bone (Musculoskeletal and connective tissue disorders) | 6 (6) — number of subjects effected: Grade 1=5 grade 2=0 grade 3=1
pain: chestwall (Skin and subcutaneous tissue disorders) | 4 (4) — number of subjects effected: Grade 1=2 grade 2=2 grade 3=0
pain:extremity (Musculoskeletal and connective tissue disorders) | 6 (6) — number of subjects effected: Grade 1=3 grade 2=2 grade 3=1
pain: headache (Nervous system disorders) | 11 (11) — number of subjects effected: Grade 1=9 grade 2=2 grade 3=0
pain:joint (Musculoskeletal and connective tissue disorders) | 9 (9) — number of subjects effected: Grade 1=4 grade 2=3 grade 3=2
pain: muscle (Musculoskeletal and connective tissue disorders) | 4 (4) — number of subjects effected: Grade 1=1 grade 2=3 grade 3=0
elevated ALT (Hepatobiliary disorders) | 5 (5) — number of subjects effected: Grade 1=4 grade 2=1 grade 3=0
elevated AST (Hepatobiliary disorders) | 4 (4) — number of subjects effected: Grade 1=2 grade 2=0 grade 3=0
hyponatremia (Investigations) | 2 (2) — number of subjects effected: Grade 1=1 grade 2=0 grade 3=1
thrombocytopenia (Investigations) | 2 (2) — number of subjects effected: Grade 1=0 grade 2=1 grade 3=1
DVT (Vascular disorders) | 2 (2) — number of subjects effected: Grade 1=0 grade 2=0 grade 3=2
edema:facial (General disorders) | 5 (5) — number of subjects effected: Grade 1=4 grade 2=1 grade 3=0
edema: extremity (General disorders) | 6 (6) — number of subjects effected: Grade 1=5 grade 2=1 grade 3=0
cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — number of subjects effected: Grade 1=0 grade 2=0 grade 3=1
rash (Skin and subcutaneous tissue disorders) | 16 (16) — number of subjects effected: Grade 1=14 grade 2=2 grade 3=0
mucositis (Skin and subcutaneous tissue disorders) | 4 (4) — number of subjects effected: Grade 1=4 grade 2=0 grade 3=0
rhinitis (General disorders) | 5 (5) — number of subjects effected: Grade 1=5 grade 2=0 grade 3=0
neuropathy sensory (Nervous system disorders) | 9 (9) — number of subjects effected: Grade 1=7 grade 2=2 grade 3=0
plueral effusion (Respiratory, thoracic and mediastinal disorders) | 16 (16) — number of subjects effected: Grade 1=5 grade 2=8 grade 3=3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No